CLINICAL TRIAL: NCT00434382
Title: Neuronale Mechanismen Der Sensorischen Reizverarbeitung in Der Narkose
Brief Title: Neuronal Mechanisms of Sensory Processing During General Anesthesia
Acronym: BEO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: C. R. Bard (Industry); German Federal Ministry of Education and Research (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BMBF 0311537
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2007-02

CONDITIONS: General Anesthesia
Keywords: auditory evoked potentials; sensory processing; monitoring; general anesthesia
MeSH Terms: interventions — Sevoflurane; Isoflurane; Desflurane; Propofol; Fentanyl; Sufentanil; Alfentanil; Remifentanil

INTERVENTIONS:
Drug: Sevoflurane
Drug: Isoflurane
Drug: Desflurane
Drug: Propofol
Drug: Fentanyl
Drug: Sufentanil
Drug: Alfentanil
Drug: Remifentanil
Device: Midlatency auditory evoked potentials

SUMMARY:
The ability of Mid Latency Auditory Evoked Potentials for a routine monitoring of sensory suppression should be evaluated during a wide spectrum of clinically common forms general anesthesia.

DETAILED DESCRIPTION:
Up to now there is no fully functional and precise technique for accurate assessment for monitoring the degree of unconsciousness during general anaesthesia. Previous studies and results obtained during the project regarding the effect of anaesthetics on single neurons and small neuronal networks indicate that it would be most promising to use a method directly correlating to the integrity of the relevant functional systems. As one goal of the project it was formulated to develop and test a new system for recording and analysis of mid latency auditory evoked potentials (MLAEP), suitable to be used in the clinical surrounding of an operation theatre. Step by step an investigational system was developed, that after obtaining legal approvement was functional in a broad spectrum of cases. In a multicenter study the including 4 clinical centres and 426 patients the reliability of the system was proved. Even under the hard conditions of the OR the apparatus was able to record the signals with sufficient reliability and precision. A clear correlation of MLAEP parameters with clinically defined states of consciousness could be identified. Differences in the effect of the used combinations of general anaesthetics and opioids were identified. An algorithm for automatic analysis of the signals was developed, to allow users with limited knowledge of interpretation of MLAEP signals to use them for monitoring anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Scheduled for elective urological, gynaecological or general surgery
* ASA status I or II
* Age 18 to 65

Exclusion Criteria:

* ASA status above II
* Operative procedures involving the neurocranium, neck or require other neurophysiologic monitoring
* Inability to communicate freely in the german language
* Major hearing deficit
* Regular centrally acting medication including drug abuse within 3 months prior to the investigation
* Participant of an other clinical investigation
* Lacking or withdrawal of written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 768
Dates: Start 2002-10; Study Completion 2003-12

PRIMARY OUTCOMES:
Intraoperative signs of inadequate anesthesia
Postoperative recall of events
MLAEP parameters

CONTACTS AND LOCATIONS:
Overall Officials: Michael AM Daunderer, M.D.,Ph.D., Principal Investigator — Klinik fuer Anaesthesiologie, Ludwig-Maximilians-Universitaet Muenchen
Locations (4):
- Germany (4):
  - Krankenhaus Friedrichshafen, Friedrichshafen
  - Klinik für Anaesthesia am Universitaetsklinikum Heidelber, Heidelberg
  - Klinik fuer Anaesthesiologie am Universitätsklinikum Schleswig Holstein, Campus Luebeck, Lübeck
  - Klinik fuer Anaesthesiologie der Ludwigs-Maximilians-Universitaet Muenchen, Munich

REFERENCES:
- [Derived] Scheller BC, Daunderer M, Pipa G. General anesthesia increases temporal precision and decreases power of the brainstem auditory-evoked response-related segments of the electroencephalogram. Anesthesiology. 2009 Aug;111(2):340-55. doi: 10.1097/ALN.0b013e3181acf7c0. PMID 19602953
- See also: homepage of the institute for medical psychology of the Ludwigs-Maximilians-University Munich — http://www.imp.med.uni-muenchen.de/index.html